CLINICAL TRIAL: NCT05625763
Title: State of Coagulation in Pre-eclampsia: Comparing Sonoclot Signature Analysis With Conventional and Specific Haemostasis Assays
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, menna nashat, assiut- elgomhoriaa, Assiut University
Other Study IDs: koshy
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: sonoclot signature analysis — Investigate the value of global hemostasis studies (Sonoclot signature analysis) in cases of pre-eclampsia and if there a correlation between it and the specific traditional assays of hemostasis.

SUMMARY:
* Detection of the presence or absence of coagulopathy in cases with pre-eclampsia.
* Investigate the value of global hemostasis studies (Sonoclot signature analysis) in cases of pre-eclampsia and if there a correlation between it and the specific traditional assays of hemostasis.

DETAILED DESCRIPTION:
Pre-eclampsia remains a major cause of morbidity and mortality in pregnant women, as well in their newborns (1). Despite intense study, preeclampsia remains poorly understood and a major cause of maternal and foetal morbidity and mortality. It's clear that vascular endothelial dysfunction, which may lead to hypertension by imbalance between vasoactive, and vasodilator agents, is an important component of this disorder. The induction of endothelial dysfunction is probably multifactorial (2). Some researchers suggested that hereditary and acquired thrombophilia has been associated with recurrent pregnancy loss and gestational vascular complications, such as early-onset pre-eclampsia and placental abruption (3). Despite it is widely known that pregnancy induces a state of hypercoagulability (4), publications failed to demonstrate a uniform pattern of pathology that can carry the association between thrombophilia and adverse pregnancy outcomes, as between factor V Leiden mutation, MTHFR C677T mutation, G20210A Prothrombin gene mutation, Anti-thrombin III deficiency, Protein C,S deficiency and other causes of thrombophilia, different researchers claimed different causes of the previously mentioned as the one responsible for maternal thrombophilia (2, 3, 5). Others claimed racial variations were associated with the state of thrombophilia (6).

Other than standard routine and specific tests, various other methods are used to record coagulation profile. One of them is estimation by sonoclot, which is a viscoelastic hemostatic assays device (7). Sonoclot have practical advantages as point-of-care device for monitoring major hemorrhage including a set of parameters that assesses a global coagulation profile and can indicate the presence of hypercoagulable state (8). Establishing correlations between Sonoclot parameters and conventional hemostasis assays could open a path of better monitoring of patients with suspected coagulopathies, and can be helpful in guiding management of preeclampsia and preventing severe maternal outcomes (7).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant pre-eclamptic patients with blood pressure > 140/90 mm hg and proteinuria > 0.39/24 hrs., with gestational age between 20-42 weeks (second & third trimester).
2. Pregnant normotensive females with no pregnancy complications and gestational age 20-42 weeks to act as controls.

Exclusion Criteria:

1. Patients with gestational age < 20 weeks (First trimester).
2. Patients in labour.
3. Patients with foetal malformations, history of chronic hypertension, diabetes mellitus, renal diseases, collagen vascular disease, anaemia, cardiovascular diseases and patients known to be thrombophilic before pregnancy (acquired or inherited).

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: * Pregnant pre-eclamptic patients with blood pressure > 140/90 mm hg and proteinuria > 0.39/24 hrs., with gestational age between 20-42 weeks (second & third trimester).
  * Pregnant normotensive females with no pregnancy complications and gestational age 20-42 weeks to act as controls.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
sonoclot signature analysis in pre-eclampsia | baseline
  Investigate the value of global hemostasis studies (Sonoclot signature analysis) in cases of pre-eclampsia and if there a correlation between it and the specific traditional assays of hemostasis.

REFERENCES:
- [Background] Lalic-Cosic S, Dopsaj V, Kovac M, Pruner I, Littmann K, Mandic-Markovic V, Mikovic Z, Antovic A. Evaluation of global haemostatic assays and fibrin structure in patients with pre-eclampsia. Int J Lab Hematol. 2020 Jun;42(3):322-330. doi: 10.1111/ijlh.13183. Epub 2020 Mar 19. PMID 32190981
- [Background] Osmanagaoglu MA, Topcuoglu K, Ozeren M, Bozkaya H. Coagulation inhibitors in preeclamptic pregnant women. Arch Gynecol Obstet. 2005 Mar;271(3):227-30. doi: 10.1007/s00404-003-0596-4. Epub 2004 Jan 21. PMID 14735372
- [Background] Greer IA, Aharon A, Brenner B, Gris JC. Coagulation and placenta-mediated complications. Rambam Maimonides Med J. 2014 Oct 29;5(4):e0034. doi: 10.5041/RMMJ.10168. eCollection 2014 Oct. PMID 25386350
- [Background] Simcox LE, Ormesher L, Tower C, Greer IA. Thrombophilia and Pregnancy Complications. Int J Mol Sci. 2015 Nov 30;16(12):28418-28. doi: 10.3390/ijms161226104. PMID 26633369
- [Background] Alfirevic Z, Roberts D, Martlew V. How strong is the association between maternal thrombophilia and adverse pregnancy outcome? A systematic review. Eur J Obstet Gynecol Reprod Biol. 2002 Feb 10;101(1):6-14. doi: 10.1016/s0301-2115(01)00496-1. PMID 11803092
- [Background] Philipp CS, Faiz AS, Beckman MG, Grant A, Bockenstedt PL, Heit JA, James AH, Kulkarni R, Manco-Johnson MJ, Moll S, Ortel TL. Differences in thrombotic risk factors in black and white women with adverse pregnancy outcome. Thromb Res. 2014 Jan;133(1):108-11. doi: 10.1016/j.thromres.2013.10.035. Epub 2013 Nov 1. PMID 24246297
- [Background] Saxena P, Bihari C, Rastogi A, Agarwal S, Anand L, Sarin SK. Sonoclot signature analysis in patients with liver disease and its correlation with conventional coagulation studies. Adv Hematol. 2013;2013:237351. doi: 10.1155/2013/237351. Epub 2013 Dec 11. PMID 24396346
- [Background] Min J, Wan P, Liu G, Yu M, Su L. Sonoclot Signature Analysis: A New Point-of-Care Testing Method for Defining Heat Stroke-Induced Coagulopathy. Int J Gen Med. 2021 Oct 20;14:6925-6933. doi: 10.2147/IJGM.S321982. eCollection 2021. PMID 34707386